CLINICAL TRIAL: NCT00741611
Title: A Randomized Controlled Trial of Radiofrequency Ablation for the Treatment of Paroxysmal Atrial Fibrillation Using the Bard High Density Mesh Ablation System (MAGELLAN)
Brief Title: Study of HD Mesh Ablation System for Treatment of Paroxysmal Atrial Fibrillation
Acronym: MAGELLAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEP-4408-2007; IDE # G070179
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesh (Experimental): Ablation with HD Mesh Ablation System
  Interventions: Device: HD Mesh Ablation System
- Drug (Active Comparator): Treatment with anti-arrhythmic drugs
  Interventions: Drug: Anti-arrhythmic drugs

INTERVENTIONS:
Device: HD Mesh Ablation System — Ablation using the HD Mesh Ablation System
  Arms: Mesh
Drug: Anti-arrhythmic drugs — 5 anti-arrhythmic drugs administered at the labeled dosage for atrial fibrillation
  Arms: Drug

SUMMARY:
This is a randomized controlled study of the Bard High Density Mesh Ablation System for treatment of paroxysmal atrial fibrillation. This study will determine if the HD Mesh Ablation System is as safe as and more effective than anti-arrhythmic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic paroxysmal atrial fibrillation who have failed at least one class I or III anti-arrhythmic drug
* Other inclusion criteria

Exclusion Criteria:

* Previous surgical or catheter ablation to treat AF
* Permanent AF
* Uncontrolled or unstable medical conditions
* Other exclusion criteria

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Harcarik, Study Director — C. R. Bard, Inc.
Locations (13):
- United States (13):
  - University of California, San Diego Medical Center, San Diego, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Heart Group, Orlando, Florida
  - Bay Heart Group, Tampa, Florida
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Northeast Cardiology Associates, Bangor, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - St. John's Medical Research Institute, Springfield, Missouri
  - Lehigh Valley Heart Specialists, Allentown, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2008 and November 2009, 44 patients were enrolled into the study. The study Sponsor made a business decision in late November 2009 to terminate the trial early; enrollment was closed at that time.
Pre-assignment Details: Of the 44 enrolled patients, a total of 36 patients were treated. Treated patients were followed for 12 months.
Groups:
- Mesh: Ablation with HD Mesh Ablation System; energy delivered to the heart tissue intended to disrupt the abnormal electrical pathways which cause atrial fibrillation to occur.
- Drug: Treatment with anti-arrhythmic drugs: treatment was selected by the Investigator and administered in accordance with the approved drug labeling using labeled doses for the atrial fibrillation indication. Per protocol, medications were limited to sotalol, flecainide, propafenone, dofetilide, and amiodarone and did not include rate control medications or calcium chanel blockers.
- Roll-ins: Investigator's first patients treated with the experimental mesh ablation system prior to the start of the study randomization.
Period: Overall Study
Arm/Group | Mesh | Drug | Roll-ins
Started | 4 | 3 | 29
Completed | 4 | 1 | 26
Not Completed | 0 | 2 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Roll-ins: Investigator's first patients treated with mesh prior to the start of the study randomization.
- Total: Total of all reporting groups
Arm/Group | Mesh | Drug | Roll-ins | Total
Number analyzed (Participants) | 4 | 3 | 29 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.18) | 66.0 (9.54) | 60.2 (9.68) | 61.2 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 9 | 11
  Male | 2 | 3 | 20 | 25
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 29 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Complications
Description: A Major Complication was defined as any adverse event that met the following criteria: 1) event was a Serious Adverse Event; 2) event was related to study device (mesh/mesh toolkit) or study procedure and 3)event was a) a cardiovascular adverse event occurring within 7 days of the procedure and/or b) a direct ablation effect adverse event occurring within 12 months of the study procedure.
Time Frame: 12 months
Population: Patients who were treated with the HD Mesh Ablation System
Measure: Number; unit: participants
Arm/Group | Mesh | Roll-ins
Number analyzed (Participants) | 4 | 29
participants | 0 | 2

2. Primary Outcome: Number of Participants With Serious Atrial Fibrillation Events
Description: Due to the early study termination and the small number of randomized patients (seven), this primary endpoint analysis (comparison of the rate of events in the mesh group to the rate in the drug group) could not be performed. Counts of events occurring in the 36 treated patients are reported by study group instead.
Time Frame: 12 months
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | Mesh | Drug | Roll-ins
Number analyzed (Participants) | 4 | 3 | 29
participants | 1 | 0 | 2

3. Primary Outcome: Number of Participants With Freedom From Symptomatic Atrial Fibrillation
Description: Due to the early termination and the enrollment of only seven randomized patients, the endpoint was not evaluable.
Time Frame: 12 months
Population: All treated patients
Arm/Group | Mesh | Drug | Roll-ins
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With the Occurrence of Pulmonary Vein Stenosis in Mesh Treated Patients.
Description: Defined as a greater than or equal to 70% diameter reduction in a pulmonary vein compared with the baseline measurement as assessed by an independent core imaging laboratory.
Time Frame: 12 months
Population: All mesh treated patients.
Measure: Number; unit: participants
Arm/Group | Mesh | Roll-ins
Number analyzed (Participants) | 4 | 29
participants | 0 | 0

5. Secondary Outcome: Number of Participants With Acute Procedural Success in Mesh Treated Patients.
Description: Acute procedural success was defined as the ability to isolate 3 of 4 pulmonary veins with the mesh ablation system alone without the need for further ablation with a distal tip catheter
Time Frame: During the mesh ablation procedure
Population: All mesh treated patients.
Measure: Number; unit: participants
Arm/Group | Mesh | Roll-ins
Number analyzed (Participants) | 4 | 29
participants | 4 | 23

ADVERSE EVENTS:
Time Frame: 12 months post procedure
Arm/Group | Mesh | Drug | Roll-ins
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 16/29
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesh (N=4) | Drug (N=3) | Roll-ins (N=29)
Prothrombin time shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 6 (7) — Note: not all 7 serious adverse events of atrial fibrillation met the predefined protocol criteria for the outcome measure of "Serious Atrial Fibrillation Events."
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Myoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Event was considered a protocol defined Major Complication; event resulted in patient death.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Event was considered a protocol defined Major Complication. A procedure was performed to remove the fluid and the event resolved.
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesh (N=4) | Drug (N=3) | Roll-ins (N=29)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 9 (9)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and enrollment of only 7 randomized patients, predefined study endpoints were not evaluable. Treated patients were followed through 12 months postprocedure and data were summarized where possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to public release at least 60 days prior to publication and that the multi-center results should be published prior to any individual site results unless the multi-center results are not published 2 years after the trial is complete. The only embargo that the sponsor can impose is on the release of confidential information.